CLINICAL TRIAL: NCT00627107
Title: Study of the ReWalk Motorized Exoskeleton Suit That Enables Individuals With Lower Limbs Impairment to Walk and to Perform Other Basic Mobility Functions.
Brief Title: A Study Testing Safety and Tolerance of the ReWalk Exoskeleton Suit
Acronym: RW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReWalk Robotics, Inc. (Industry)
Responsible Party: Dr. Gabi Zeilig, Head of the Neurological Rehabilitation Department (PI), Sheba Medical center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RW-002
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Paraplegia; SCI
Keywords: ReWalk, Paraplegia, SCI
MeSH Terms: conditions — Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): A group of paraplegics.
  Interventions: Device: ReWalk - a motorized exoskeleton suit

INTERVENTIONS:
Device: ReWalk - a motorized exoskeleton suit — The subject will wear the ReWalk suit and have training sessions for walking with the device.
  Other Names: Exoskeleton suit

SUMMARY:
The ReWalk enables people with lower limb disabilities to carry out routine ambulatory functions (stand, walk, climb stairs etc.). It can be used by people with disabilities such as spinal cord injury, brain injury, stroke, multiple sclerosis, cerebral palsy and other severe walking impairments. The device promises to restore the dignity of disabled persons, enabling them to work and improve their general health and quality of life, as well as significantly reduce medical and other related expenses.

DETAILED DESCRIPTION:
The ReWalk comprises light wearable brace support suit, which integrates DC motors at the joints, rechargeable batteries, an array of sensors and a computer-based control system. It is snugly fitted on the body and worn underneath the clothing, if desired. ReWalk is a new realization of the Powered Exoskeleton concept, first tried about fifty years ago with no success. Employing an innovative, non-robotic design approach, it uniquely matches the user's capabilities with the control mechanisms. Upper-body movements of the user are detected and used to initiate and maintain walking processes. User stability and safety during ambulation is secured by concurrent use of safety aids such as crutches for walking and railing for stairs.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (at least 6 months after injury) complete cervical(C7-8) or thoracic (T1-T12) spinal cord injury
* Age between 18-55
* Male and non-pregnant non-lactating female
* Regular use of RGO or bing able to stand up using a device (e.g. EasyStand)
* under 100 kg and between 155-200 cm of height

Exclusion Criteria:

* History of severe neurological injuries other than SCI (MS, CP, ALS, TBI etc)
* Severe concurrent medical diseases: infections, heart or lung, pressure sores
* Unstable spine or unhealed limbs or pelvic fractures
* Psychiatric or cognitive situations that may interfere with the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Observation and subject feedback | 3 months

SECONDARY OUTCOMES:
subject tolerance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabi Zeilig, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Neurological Rehabilitation Department, Tel Litwinsky, Israel